CLINICAL TRIAL: NCT04631861
Title: Physical Activity and the Risk of COVID-19 Infection and Mortality
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hyuk Cho, Clinical assistant professor, Wonju Severance Christian Hospital
Other Study IDs: 2020AN0292
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Covid19
Keywords: Physical activity
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Currently, there is no cure for COVID-19, except for supportive treatments. Quarantine for a defined period is the best option to reduce the spread of COVID-19. Physical activity has been shown to reduce the risk of serious community-acquired infections. However, it remains unanswered is whether physical activity has protective effects against SARS-CoV-2 infection and COVID-19 related mortality. This study aimed to examine the association of PA with the morbidity and mortality of COVID-19 infection in the entire South Korean population.

ELIGIBILITY:
Inclusion Criteria:

* all Koreans who tested positive for SARS-CoV-2
* more than 18 years old
* who underwent public health screening between 2014 and 2017

Exclusion Criteria:

* missing values about physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Korean nationwide COVID-19 study was a retrospective, nationwide study including all Koreans who tested positive for SARS-CoV-2, aimed at evaluating the characteristics and outcomes of patients with COVID-19. Case patients were defined as individuals over 18 years old with positive results for the SARS-CoV-2 test. For every case patient, we selected up to 20 random controls from the target population who underwent the national health screening.
Sampling Method: Probability Sample
Enrollment: 132069 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 positivity rate (%) | 7 years
  The SARS-CoV-2 infection was confirmed using the real-time reverse transcriptase polymerase chain reaction of pharyngeal and nasal swab samples, in accordance with the WHO recommendations
COVID-19 related mortality rate (%) | 7 years
  The COVID-19 related mortality was defined as the termination of isolation due to death.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hyuk Cho, Principal Investigator — Yonsei Wonju Christian Hospital

IPD SHARING:
Plan to Share IPD: No
The present study are not publicly accessible due to Korean personal information projection act.

REFERENCES:
- [Result] Phelan AL, Katz R, Gostin LO. The Novel Coronavirus Originating in Wuhan, China: Challenges for Global Health Governance. JAMA. 2020 Feb 25;323(8):709-710. doi: 10.1001/jama.2020.1097. No abstract available. PMID 31999307
- [Result] Cucinotta D, Vanelli M. WHO Declares COVID-19 a Pandemic. Acta Biomed. 2020 Mar 19;91(1):157-160. doi: 10.23750/abm.v91i1.9397. PMID 32191675
- [Result] Kim DW, Byeon KH, Kim J, Cho KD, Lee N. The Correlation of Comorbidities on the Mortality in Patients with COVID-19: an Observational Study Based on the Korean National Health Insurance Big Data. J Korean Med Sci. 2020 Jul 6;35(26):e243. doi: 10.3346/jkms.2020.35.e243. PMID 32627443
- [Result] Hamer M, Kivimaki M, Gale CR, Batty GD. Lifestyle risk factors, inflammatory mechanisms, and COVID-19 hospitalization: A community-based cohort study of 387,109 adults in UK. Brain Behav Immun. 2020 Jul;87:184-187. doi: 10.1016/j.bbi.2020.05.059. Epub 2020 May 23. PMID 32454138